CLINICAL TRIAL: NCT02440685
Title: A Phase 1/2, Open-Label, Uncontrolled, Multiple Dose Escalation, Cohort Expansion Study To Evaluate The Safety, Tolerability, Pharmacokinetics And Preliminary Efficacy Of ASN002 In Relapsed/Refractory Lymphoma, Myelofibrosis, Chronic Lymphocytic Leukemia, And Advanced Solid Tumors
Brief Title: A Phase 1/2 Study To Evaluate ASN002 In Relapsed/Refractory Lymphoma And Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: Asana BioSciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASN002-101
Record Dates: First submitted 2015-05-05; First posted 2015-05-12 (Estimated); Results first posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, Follicular; Cancer; Neoplasm; Tumor; Lymphoma, Malignant; Lymphoma, B-cell; Lymphoma, Non-Hodgkin; B-Cell Chronic Lymphocytic Leukemia; B-Cell Leukemia, Chronic; B-Lymphocytic Leukemia, Chronic; Chronic Lymphocytic Leukemia; Leukemia, Lymphocytic, Chronic; Leukemia, Lymphocytic, Chronic, B Cell; Myelofibrosis; Chronic Idiopathic Myelofibrosis; Idiopathic Myelofibrosis; Lymphoma, T Cell, Peripheral; Peripheral T-Cell Lymphoma; T-Cell Lymphoma, Peripheral
Keywords: DLBCL; FL; MCL; PTCL; MF; CLL
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, Follicular; Neoplasms; Lymphoma; Lymphoma, B-Cell; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Primary Myelofibrosis; Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Intervention Model Description: Study terminated early so no all groups per protocol were conducted
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A ASN002 Dose Escalation (Experimental): Multiple ascending doses of ASN002 will be administered to determine the maximum tolerated dose (MTD). Arm Closed
  Interventions: Drug: ASN002 Dose Escalation
- Part B ASN002 Recommended dose (RD) (Experimental): ASN002 administered at the recommended dose
  Interventions: Drug: ASN002 RD

INTERVENTIONS:
Drug: ASN002 Dose Escalation — Multiple ascending doses of ASN002 assigned by cohort
  Arms: Part A ASN002 Dose Escalation
Drug: ASN002 RD — Recommended dose of ASN002 from Part A
  Arms: Part B ASN002 Recommended dose (RD)

SUMMARY:
This study is a dose escalation, and cohort expansion study in subjects with advanced cancer for which no standard therapy exists. Subjects must have received prior treatment for cancer that has not worked, or has stopped working.

DETAILED DESCRIPTION:
The study will be conducted in two parts. Part A is a dose escalation study to determine a safe and tolerable dose of ASN002 for subjects with relapsed or refractory lymphoma, or advanced solid tumors. Part A will also characterize the pharmacokinetics and pharmacodynamics of ASN002 through blood sampling. Subjects in Part B will enroll subjects with four types of lymphoma Diffuse Large B-cell Lymphoma (DLBCL), Follicular Lymphoma (FL), Mantle Cell Lymphoma (MCL) and Peripheral T-cell lymphoma (PTCL). Additional groups of subjects with Myelofibrosis (MF) and Chronic Lymphocytic Leukemia (CLL) will be enrolled. Subjects will be treated with the highest safe and tolerable dose determined in Part A of the study to determine preliminary efficacy. Subjects may continue to receive ASN002 for up to 1 year in the absence of severe side effects or disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to any study-related procedure being performed;
* Male or female subjects at least 18 years of age at the time of consent;
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2;
* Recovered from the reversible effects of prior antineoplastic therapy (with the exception of alopecia and Grade 1 neuropathy).
* Screening blood counts of the following: Absolute neutrophil count ≥ 1000/μL, Platelets ≥ 75,000/μL, Hemoglobin ≥ 8 g/dL (with transfusion support);
* Screening chemistry values of the following: Alanine aminotransferase (ALT) and aspartate transaminase (AST) ≤ 3.0 × upper limit of the normal (ULN), total bilirubin ≤ 1.5 × ULN, Creatinine ≤ 1.5 × ULN;
* At screening, life expectancy of at least 3 months;
* Subject is willing and able to comply with all protocol required visits and assessments;
* Male and female subjects of child-bearing potential must agree to use medically acceptable methods of birth control throughout the study and for thirty (30) days after the last dose of study medication.
* (Part A only) Histologically or cytologically confirmed metastatic and/or advanced solid tumors or lymphomas for which no standard therapy exists, or who are not eligible for standard treatment. Subjects must have received at least one prior therapy for their malignancy;
* (Part B only) Histologically confirmed DLBCL/MCL/FL/PTCL/MF/CLL on the basis of excisional lymph node or extranodal tissue biopsy; diagnosis of relapsed/refractory disease defined as 1) recurrence of disease after a Complete Response (CR), or 2) Partial Response (PR), Stable Disease (SD) at completion of treatment regimen preceding entry into study, subjects must not be candidates for standard therapy, subjects who have not received Stem Cell Translplant (SCT) must be ineligible to receive SCT.

Exclusion Criteria

* Have received prior chemotherapy regimens within 4 weeks of Day 1;
* Have received prior treatment with monoclonal antibodies within 6 weeks of first dose of Day 1;
* Have had major surgery within 30 days prior to the start of Day 1;
* Received any investigational treatment within 4 weeks prior to the start of study medication;
* Have had an infection requiring the use of parenteral antibiotics within 14 days prior to the start of Day 1;
* Have known central nervous system metastasis or Central Nervous System lymphoma;
* Is receiving high dose corticosteroids (>10 mg prednisone daily or equivalent);
* Has known bleeding diathesis that would be a safety risk;
* Has a history of other malignancy within the 3 years prior to screening, except adequately treated basal cell or squamous cell carcinoma of the skin, or carcinoma in-situ;
* Has difficulty swallowing medications, or known history of malabsorption syndrome;
* Has a serious concurrent medical condition, such as: congestive heart failure New York Heart Association (NYHA) class III or IV or uncontrolled hypertension at screening, 12-Lead electrocardiogram (ECG) abnormalities considered by the investigator to be clinically significant including myocardial infarction, angioplasty, or cardiac stent placement within the last 6 months, HIV infection, known Hepatitis B or C infection. Subjects at high risk for Hepatitis B or C infection should have serology testing to rule out infection, a medical condition requiring the therapeutic use of anticoagulants.
* Known hypersensitivity to ASN002 or its excipients;
* Prior participation, i.e., receipt of study medication, in this study;
* Any condition that, in the opinion of the investigator, would impair the subject's ability to comply with study procedures;
* Female subjects that are pregnant or lactating.
* Part B only: Prior treatment with SYK or Janus Kinase (JAK) inhibitors, except MF subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Niranjan Rao, PhD, Study Director — Asana BioSciences
Locations (14):
- United States (12):
  - Arizona Oncology, Tempe, Arizona
  - University of California, San Francisco, San Francisco, California
  - Winship Cancer Institute - Emory, Atlanta, Georgia
  - University of Michigan, Ann Arbor, Michigan
  - START - Midwest, Grand Rapids, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Gabrail Cancer Center, Canton, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
- Argentina (2):
  - Hospital Universitario Austral, Buenos Aires, Derqui, Pilar
  - Instituto Alexander Fleming, Buenos Aires

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 10 mg BID: ASN002 Dose 10 mg BID
- 20 mg BID: ASN002 20 mg BID
- 30 mg BID: ASN002 30 mg BID
- 40 mg BID: ASN002 40 mg BID
- 50 mg BID: ASN002 50 mg BID
- 75 mg BID: ASN002 75 mg BID
- 100 mg BID: ASN002 100 mg BID
- 80 mg QD: ASN002 80 mg QD
- 120 mg QD: ASN002 120 mg QD
Period: Overall Study
Arm/Group | 10 mg BID | 20 mg BID | 30 mg BID | 40 mg BID | 50 mg BID | 75 mg BID | 100 mg BID | 80 mg QD | 120 mg QD
Started | 3 | 4 | 3 | 4 | 7 | 15 | 5 | 7 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 4 | 3 | 4 | 7 | 15 | 5 | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- 10 mg BID: ASN002 10 mg BID
- Total: Total of all reporting groups
Arm/Group | 10 mg BID | 20 mg BID | 30 mg BID | 40 mg BID | 50 mg BID | 75 mg BID | 100 mg BID | 80 mg QD | 120 mg QD | Total
Number analyzed (Participants) | 3 | 4 | 3 | 4 | 7 | 15 | 5 | 7 | 3 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (19.31) | 67.5 (9.47) | 66.3 (5.51) | 62.0 (6.68) | 62.9 (20.39) | 65.1 (9.92) | 63.2 (13.81) | 65.6 (10.33) | 74.0 (7.00) | 65.2 (11.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 4 | 4 | 3 | 1 | 4 | 0 | 20
  Male | 2 | 3 | 1 | 0 | 3 | 12 | 4 | 3 | 3 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 0 | 3 | 3 | 1 | 2 | 0 | 12
  Not Hispanic or Latino | 2 | 4 | 1 | 4 | 4 | 12 | 4 | 5 | 3 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 3 | 4 | 3 | 4 | 7 | 15 | 5 | 6 | 3 | 50
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disease Characteristic [Count of Participants; unit: Participants]
  Lymphoma | 0 | 1 | 0 | 2 | 4 | 11 | 2 | 4 | 1 | 25
  Solid tumor | 3 | 3 | 3 | 2 | 3 | 2 | 3 | 3 | 2 | 24
  Myelofibrosis | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Due to the early termination of the study, data for efficacy endpoints were insufficient for the planned efficacy analyses.
Time Frame: First 29 days
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg BID | 20 mg BID | 30 mg BID | 40 mg BID | 50 mg BID | 75 mg BID | 100 mg BID | 80 mg QD | 120 mg QD
Number analyzed (Participants) | 3 | 4 | 3 | 4 | 7 | 15 | 5 | 7 | 3
Participants
  Not evaluable | 0 | 1 | 0 | 2 | 2 | 12 | 3 | 1 | 0
  Complete response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial response | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Stable disease | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 2 | 1
  Progressive disease | 3 | 1 | 2 | 2 | 4 | 1 | 2 | 4 | 1

ADVERSE EVENTS:
Time Frame: Days of duration ranged from 4 days to 280 days before early termination of the study
Arm/Group | 10 mg BID | 20 mg BID | 30 mg BID | 40 mg BID | 50 mg BID | 75 mg BID | 100 mg BID | 80 mg QD | 120 mg QD
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/4 | 0/3 | 1/4 | 2/7 | 6/15 | 2/5 | 0/7 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/4 | 0/3 | 2/4 | 5/7 | 10/15 | 4/5 | 4/7 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 2/3 | 4/4 | 6/7 | 14/15 | 5/5 | 7/7 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 10 mg BID (N=3) | 20 mg BID (N=4) | 30 mg BID (N=3) | 40 mg BID (N=4) | 50 mg BID (N=7) | 75 mg BID (N=15) | 100 mg BID (N=5) | 80 mg QD (N=7) | 120 mg QD (N=3)
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 10 mg BID (N=3) | 20 mg BID (N=4) | 30 mg BID (N=3) | 40 mg BID (N=4) | 50 mg BID (N=7) | 75 mg BID (N=15) | 100 mg BID (N=5) | 80 mg QD (N=7) | 120 mg QD (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 3 | 5 | 0 | 3 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 5 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 4 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 2 | 6 | 0 | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0
Chills (General disorders) | 1 | 0 | 0 | 1 | 1 | 2 | 2 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 0 | 1 | 1 | 4 | 2 | 1 | 2
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 3 | 3
Headache (Nervous system disorders) | 2 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Oral Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0
Blood creatinine increase (Investigations) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0
Arthralagia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-05-24): https://cdn.clinicaltrials.gov/large-docs/85/NCT02440685/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-24): https://cdn.clinicaltrials.gov/large-docs/85/NCT02440685/SAP_001.pdf